CLINICAL TRIAL: NCT06324591
Title: Multicentre Observational Cohort Study in Newly Diagnosed Crohn's Disease Patients Aimed at Identifying Intestinal Microbial Profiles Correlated With Low and High Risk of Severe Disease Course
Brief Title: Observational Prospective Study to Identify Intestinal Microbial Profiles in Newly Diagnosed Crohn's Disease Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Paolo Lionetti, Principal Investigator, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RISKCROHNBIOM
Record Dates: First submitted 2024-02-22; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with Chron's Disease (Other): Only patient with Crohn's Disease
  Interventions: Other: Collection biological sample and analysis

INTERVENTIONS:
Other: Collection biological sample and analysis — collection of a stool sample collected at clinical practice check-ups during the first year after diagnosis of Crohn's disease. This is followed by the evaluation of clinical, laboratory and instrumental data at the time of diagnosis

SUMMARY:
Crohn's disease (CD), a chronic inflammatory disease affecting the intestine, is characterised by a relapsing course. In 25% of cases, the onset of this disease occurs in childhood. Relevant studies have provided evidence of a key role of gut microbial communities (the microbiota) in triggering or maintaining active gut inflammation, pointing to gut dysbiosis as the main event disrupting the balance of microbial communities Recent evidence suggests that, in addition to the bacterial component, the commensal fungal component also plays a crucial role in CD.

The purpose of this prospective, longitudinal, study is to characterise the composition of intestinal bacterial and fungal communities in patients 6-18 years newly diagnosed with Crohn Disease in order to identify a possible association of specific faecal microbial profiles with a severe or mild-to-moderate disease course.

ELIGIBILITY:
Inclusion Criteria:

* Children/young people aged between 6 and 18 years with newly diagnosed CM according to recognised diagnostic criteria
* Obtaining informed consent

Exclusion Criteria:

* Refusal to participate in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Modifications in alpha and beta diversity of stool microbiome profile in patients with different phases of disease course (at diagnosis, remission and after one year of mantainance therapy) | 3 years after beginning of the study
  Detection of differences in alpha and beta diversity in stool microbiome in various phases of disease course, at diagnosis, remission and after one year of mantainance therapy

SECONDARY OUTCOMES:
Differences intestinal alpha and beta diversity, microbiome richness and composition between patients at high risk and patients at low risk | 3 years after beginning of the study
  Differences intestinal alpha and beta diversity, microbiome richness and composition between patients at high risk and patients at low risk
Indentification of different patterns of intestinal microbiome as a potential biomarker for high and low risk stratification | 3 years after beginning of the study
  Indentification of different patterns of intestinal microbiome (alpha and beta diversity, microbial richness and relative abundance of microbial species) as a potential biomarker for high and low risk patients

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Lionetti, Principal Investigator — Meyer Children's Hospital IRCCS
Locations (3):
- Medical University of Graz-Educational center for Paediatric Gastroenterology, Hepatology and Nutrition, Department of Paediatrics and adolescence medicine, Graz, Austria
- Italy (2):
  - Ospedale Maggiore-Azienda Usl Di Bologna, Bologna
  - Meyer Children's Hospital IRCCS, Florence